CLINICAL TRIAL: NCT01610115
Title: Serial HBV DNA Levels During Pregnancy in Patients With Chronic Hepatitis B: a Prospective Observational Follow-up Study
Brief Title: HBV DNA Levels During Pregnancy in Chronic Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Cheng Chen, Yi-Cheng Chen, Chang Gung Memorial Hospital
Other Study IDs: HBV-P-01
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Hepatitis B; Pregnancy
Keywords: Pregnancy
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To elucidate the natural course of chronic hepatitis B by serial HBV DNA and alanine aminotransferase (ALT) levels during pregnancy

DETAILED DESCRIPTION:
This is a prospective observational follow-up study in a single center.

Number of patients: It is estimated to enroll 100 patients in Taiwan.

Population:

Female patients with pregnancy confirmed, at least 20 years of age diagnosed with chronic hepatitis B. The patients are able to communicate well, provide informed consent and willing to participate in the entire study.

Inclusion criteria:

Patients must meet all of the following criteria

1. Documented chronic hepatitis B defined by clinical history compatible with chronic hepatitis B and detectable serum HBsAg
2. Female 20 years of age with confirmed pregnancy
3. Willing and able to comply with all the requirements in the observational followup study
4. Willing and able to provide written informed consent to participate in the study

Exclusion criteria:

Patients will be excluded from the study for any of the following reasons:

1. Concurrent infection with hepatitis C virus (HCV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV)
2. One or more known primary or secondary causes of liver disease other than hepatitis B (e.g., alcoholism, non-alcoholic steatohepatitis, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease).
3. Any other concurrent medical or psychosocial condition likely to preclude compliance with the schedule of evaluations in the protocol or likely to confound the efficacy or safety observations of the study.
4. Enrolled or planning to enroll in another clinical trial of an investigational agent while participating in this study.
5. Patients with antiviral therapy to chronic hepatitis B

ELIGIBILITY:
Inclusion Criteria:

1. Documented chronic hepatitis B defined by clinical history compatible with chronic hepatitis B and detectable serum HBsAg
2. Female 20 years of age with confirmed pregnancy
3. Willing and able to comply with all the requirements in the observational follow-up study
4. Willing and able to provide written informed consent to participate in the study

Exclusion Criteria:

1. Concurrent infection with hepatitis C virus (HCV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV)
2. One or more known primary or secondary causes of liver disease other than hepatitis B (e.g., alcoholism, non-alcoholic steatohepatitis, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease).
3. Any other concurrent medical or psychosocial condition likely to preclude compliance with the schedule of evaluations in the protocol or likely to confound the efficacy or safety observations of the study.
4. Enrolled or planning to enroll in another clinical trial of an investigational agent while participating in this study.
5. Patients with antiviral therapy to chronic hepatitis B

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Documented chronic hepatitis B defined by clinical history compatible with chronic hepatitis B and detectable serum HBsAg
  2. Female 20 years of age with confirmed pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Cheng Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan